CLINICAL TRIAL: NCT01150422
Title: The Acceptability and Feasibility of an Alternative to a Routine Follow-up Visit After Medical Abortion in Vietnam
Brief Title: The Acceptability and Feasibility of an Alternative to Routine Follow-up Visit After Medical Abortion in Vietnam
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Hillary Bracken, Gynuity Health Projects
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 6.4
Record Dates: First submitted 2010-05-07; First posted 2010-06-25 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2011-04

CONDITIONS: Medical Abortion
Keywords: medical abortion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of care for post medical abortion follow-up (No Intervention): Standard of care includes a routine hospital visit two weeks after mifepristone administration. At the hospital visit, the woman will undergo a bimanual and vaginal ultrasound examination. In the event the woman fails to return for the follow-up visit, each hospital will follow their standard procedure for contacting women who fail to attend their follow-up visit, i.e. three efforts to contact the woman. Form 2a will document the results of any clinical examinations, any additional medical abortion-related care given and the abortion outcome. At the follow-up visit, women will also be asked about the acceptability of current medical abortion follow-up procedures and their future preferences.
- Alternative follow-up (Active Comparator): At their first clinic visit, women will be asked to provide their phone number for contact purposes. Women will also be asked to complete a semi-quantitative pregnancy test in the clinic and the results of the test will be noted on a study form. After mifepristone administration, women will be provided with a second semi-quantitative pregnancy test and a self-administered checklist.
  Women will be instructed to complete the checklist and perform the pregnancy test at home on an assigned date two weeks after mifepristone administration. The checklist will indicate that if the woman answers "yes" to any of the questions, then she should return to the clinic for a follow-up visit. On the assigned date, women will also be contacted by phone by the clinic staff. Women will be asked to confirm whether they completed the pregnancy test and checklist and asked to report on the results of both tests.
  Interventions: Other: Alternative follow-up

INTERVENTIONS:
Other: Alternative follow-up — After mifepristone administration, women will be provided with a second semi-quantitative pregnancy test and a self-administered checklist. Women will be instructed to complete the checklist and perform the pregnancy test at home on an assigned data two weeks after mifepristone administration. On the assigned date, women will also be contacted by phone by the clinic staff. Women will be asked to confirm whether they completed the pregnancy test and checklist and asked to report on the results of both tests. Provider will review the women's responses to the checklist and confirm whether, based on the woman's responses, she should return for a follow up visit. During the follow-up phone call, women will also be asked about the satisfaction and acceptability of the alternative follow-up procedure.
  Arms: Alternative follow-up

SUMMARY:
This trial will compare the efficacy and acceptability of post-medical abortion follow-up by assigning women to either 1) alternative follow-up via routine semi-quantitative pregnancy test and a self-administered follow-up questionnaire, or 2) the standard of care: a routine follow-up visit including a bimanual exam and vaginal ultrasound.

The goal of the study is to provide answers to the following questions:

1. Is a follow-up protocol that employs a self-administered questionnaire and at home use of a semi-quantitative pregnancy test effective at identifying women with ongoing pregnancies?
2. Is an innovative follow-up protocol more acceptable to women and providers than the current standard of care?
3. Is an innovative follow-up protocol feasible to implement in abortion services in Vietnam?

ELIGIBILITY:
Inclusion Criteria:

* Reproductive age women seeking medical abortion services
* Intrauterine pregnancy less than or equal to 63 days gestation on the day of mifepristone administration
* Hold a working, personal phone number
* be willing and able to sign consent forms and agree to comply with study procedures

Exclusion Criteria:

* Pregnancy greater than 63 days gestation on the day of mifepristone administration

Ages: 13 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1500 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Continued, ongoing pregnancy | 9 months

SECONDARY OUTCOMES:
percentage of women who return for follow-up | 9 months
percentage of women receiving other treatment for ongoing pregnancy | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Nguyen Thi Nhu Ngoc, MD, MSc, Principal Investigator — Center for Research and Consultancy in Reproductive Health
Locations (4):
- Vietnam (4):
  - Hanoi Ob-Gyn Hospital, Hanoi
  - National Ob-Gyn Hospital, Hanoi
  - HocMon District Hospital, Ho Chi Minh City
  - Hung Vuong Hospital, Ho Chi Minh City

REFERENCES:
- [Derived] Ngoc NTN, Bracken H, Blum J, Nga NTB, Minh NH, van Nhang N, Lynd K, Winikoff B, Blumenthal PD. Acceptability and feasibility of phone follow-up after early medical abortion in Vietnam: a randomized controlled trial. Obstet Gynecol. 2014 Jan;123(1):88-95. doi: 10.1097/AOG.0000000000000050. PMID 24463668